CLINICAL TRIAL: NCT05064709
Title: Assessment of Implantable CCM in the Heart Failure Group With Higher Ejection Fraction
Brief Title: Assessment of CCM in HF With Higher Ejection Fraction
Acronym: AIM HIGHer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA_CP_340
Record Dates: First submitted 2021-09-21; First posted 2021-10-01 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mid Range Ejection Fraction; Heart Failure With Moderately Reduced Ejection Fraction; Diastolic Heart Failure
Keywords: HFpEF; Heart failure; CCM; CCM therapy; cardiac contractility modulation; symptomatic heart failure; left ventricular ejection fraction; LVEF; Optimizer; Optimizer Smart Mini; Quality of Life
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Intervention Model Description: Multicenter, multi-national, randomized, quadruple-blind, sham controlled, 2-part, embedded IDE clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: In addition to the subject, the entire site research team, the implanting physician, the Clinical Events Committee (CEC), and the clinical study monitors will all be blinded to the treatment assignment. Site research staff and Impulse Dynamics monitoring personnel will not have viewing rights to the randomization assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CCM Group (CCM ON) (Experimental): CCM therapy will be turned on in 2/3 of the subjects for the entire duration of the study.
  Interventions: Device: Cardiac Contractility Modulation Therapy via OPTIMIZER™ Smart Mini System
- Sham Group (CCM OFF) (Sham Comparator): CCM therapy will be turned off in 1/3 of the subjects for the first 18 months of the study. After 18 months, CCM therapy will be turned on for the rest of the study duration.
  Interventions: Device: OPTIMIZER™ Smart Mini System

INTERVENTIONS:
Device: Cardiac Contractility Modulation Therapy via OPTIMIZER™ Smart Mini System — The OPTIMIZER™ Smart Mini System will be implanted and CCM will be programmed ON for the first 18 months (blinded phase). CCM therapy will be programmed to deliver 7 one-hour phases of CCM therapy that are distributed equally over every 24-hour period. CCM will remain on following completion of the 18-month visit.
  Other Names: CCM Group (CCM ON)
  Arms: CCM Group (CCM ON)
Device: OPTIMIZER™ Smart Mini System — The OPTIMIZER™ Smart Mini System will be implanted and CCM will be programmed OFF for the first 18 months (blinded phase). CCM will be turned on following completion of the 18-month visit.
  Other Names: Sham Group (CCM OFF)
  Arms: Sham Group (CCM OFF)

SUMMARY:
The AIM HIGHer Clinical Trial will evaluate the safety and efficacy of Cardiac Contractility Modulation (CCM) therapy in patients with heart failure with LVEF ≥40% and ≤70%.

DETAILED DESCRIPTION:
The AIM HIGHer Clinical Trial is a prospective, multi-center, randomized, quadruple-blind, sham-controlled, two-part embedded trial of the safety and efficacy of CCM therapy delivered via the OPTIMIZER Smart Mini System in subjects with heart failure and an LVEF ≥40% and ≤70%. Subjects will be enrolled at approximately 150 sites in the US and 75 sites OUS.

All subjects will undergo screening and baseline testing; all eligible subjects will be implanted with the Optimizer System. Subjects will be randomized in a 2:1 ratio to either CCM ON (CCM group) or to CCM OFF (Sham group). The trial will be blinded to the treatment assignment of the device for 18-months. Subjects in the Sham group will have CCM turned ON after completion of the 18-month study visit. Subjects enrolled during Part I (450 subjects) of the trial will continue follow-up through the end of Part II (up to an additional 1,050) and contribute data to both parts of the trial. Each part of the trial is distinguished by a separate scientific purpose. The specific purpose of each part is:

Part I - Establish safety and effectiveness based on functional capacity and health status.

Part II - Establish safety and effectiveness based on clinical outcome data.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent form;
2. Male or non-pregnant female, 18 years or older;
3. Diagnosed with symptomatic heart failure;
4. LVEF ≥40 and ≤70% (as assessed by site echo);
5. A. Heart failure hospitalization within 12 months prior to study consent OR an urgent heart failure visit requiring IV therapy within 6 months prior to study consent OR B. If there is no heart failure hospitalization within 12 months prior to study consent OR an urgent heart failure visit requiring IV therapy within 6 months prior to study consent, an elevated BMI-adjusted natriuretic peptide value must be achieved (Refer to Table 1 in Section 9.2.6)
6. Subjects must meet one of the following conditions:

   * Have stable, scheduled oral loop diuretic treatment (not just PRN) for a minimum of 30 days before providing study consent unless there is a documented allergy or intolerance.
   * Eligibility for enrollment is maintained for patients on an SGLT2 inhibitor without prescribed concurrent standing loop diuretic therapy if investigators provide instructions for a flexible PRN diuretic regimen (deemed appropriate by the clinician in response to symptoms or weight gain) Note: Stable is defined as no more than a 100% increase or 50% decrease in dose within the last 30 days. A one-time hold of diuretic dosing for 24 hours during the 30-day period is allowed and not an exclusionary event.

Exclusion Criteria:

1. Resting ventricular rate <50 or >110 bpm;
2. Resting systolic blood pressure <100 or ≥160 mmHg;
3. BMI greater than 46
4. Any severe valvular stenotic disease or any severe valvular regurgitation;
5. Mechanical tricuspid valve;
6. Complex congenital heart disease;
7. Exercise tolerance limited by a condition other than heart failure that, in the opinion of the investigator, contributes significantly to the primary symptoms of shortness of breath and/or exercise intolerance;
8. Unable to walk at least 100 meters or walks more than 450 meters during a 6MWT;
9. A KCCQ CCS score higher than 85;
10. Hypertrophic, infiltrative/restrictive or inflammatory cardiomyopathy;
11. Unstable angina pectoris within 30 days prior to study consent;
12. Acute, decompensated heart failure requiring IV therapy or ultrafiltration within 30 days prior to consent, in the hospital or an outpatient setting;
13. Receiving cardiac resynchronization therapy (CRT); NOTE: Subjects with active/ongoing cardiac resynchronization therapy (CRT) implanted more than one year ago are eligible for inclusion if they are currently classified as NYHA class III or higher.
14. Scheduled for a cardiac surgery or a percutaneous cardiac intervention (PCI) or have undergone cardiac surgery within 90 days or a PCI procedure within 30 days prior to study consent;
15. Myocardial infarction within 90 days prior to study consent;
16. Prior heart transplant or ventricular assist device;
17. Planning to become pregnant during the study;
18. Dialysis (permanent) or GFR <15 ml/min/1.73m2;
19. Participating in another investigational drug or device study that may interfere with the interpretation of study data;
20. Currently undergoing active chemotherapeutic and/or radiation treatment for cancer or has a history of chemotherapy during the 2-year period prior to study consent;
21. Expected lifespan of less than 18 months from time of study consent;
22. Unable to follow through study protocol for any reasons in the investigator's judgement.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Part 1 Efficacy Endpoint - Change in 6-minute walk distance (6MWD) from baseline to 6 months. | 6 months
  Demonstrate that CCM therapy improves functional capacity in subjects with symptomatic heart failure with LVEF ≥40% and ≤70%. Compare the changes in functional capacity, as measured by the 6-minute walk distance (6MWD), from baseline to 6-months following the randomization date between the two study groups.
Part 1 Efficacy Endpoint - Change in the health status from baseline to 6 months as assessed by the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ CSS). | 6 months
  Demonstrate that CCM therapy improves health status in subjects with symptomatic heart failure with LVEF ≥40% and ≤60%. Compare the changes in health status, as measured by the KCCQ CSS, from baseline to 6-months following the randomization date between the two study groups.
Part 1 Safety Endpoint - The incidence of Optimizer device- or procedure-related complications within the first 12 months after implant | 12 months
  Compare the composite incidence of Optimizer device-related and procedure-related SAEs (complications) for available data collected from implant to 12 months after the Optimizer implantation procedure to a performance goal of 75% free of complications.
Part 2 Endpoint - The hierarchical composite of mortality, morbidity, and health status outcomes (KCCQ CSS). | 18 months
  Demonstrate that CCM therapy improves a composite endpoint of cardiovascular mortality at 18-months, heart failure hospitalizations at 18-months, urgent heart failure visits requiring IV diuretics at 18-months and the Kansas City Cardiomyopathy Questionnaire Clinical Summary Score (KCCQ CSS) at 12-months. Comparison of a hierarchical composite endpoint between the two study groups will be based on the Finkelstein-Schoenfeld global rank method.

CONTACTS AND LOCATIONS:
Overall Officials: Javed Butler, MD, MPH, MBA, Principal Investigator — Baylor Scott and White Research Institute, Dallas, Texas; Oussama Wazni, MD, MBA, Principal Investigator — Department of Cardiovascular Medicine, Cleveland Clinic, Cleveland, Ohio, USA
Locations (111):
- United States (111):
  - Grandview Medical Group Research, LLC, Birmingham, Alabama
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - CardioVascular Associates of Mesa, Mesa, Arizona
  - Chan Heart Rhythm Institute, Mesa, Arizona
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Banner Health- Phoenix, Phoenix, Arizona
  - Arizona Heart Rhythm, Phoenix, Arizona
  - Cardiovascular Consultants, Ltd, Phoenix, Arizona
  - HonorHealth, Scottsdale, Arizona
  - Pima Heart and Vascular, Tuscon, Arizona
  - John Muir Health, Concord, California
  - Northbay Heart and Vascular, Fairfield, California
  - University of California San Diego, La Jolla, California
  - USC Keck School of Medicine, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Valley Clinical Trials Pasadena, Northridge, California
  - Valley Clinical Trials- Northridge, Northridge, California
  - Sequoia Hospital, Redwood City, California
  - University of California Davis Health, Sacramento, California
  - University of California, San Francisco, San Francisco, California
  - Nuvance Health - Danbury Hospital, Danbury, Connecticut
  - Hartford Healthcare, Hartford, Connecticut
  - HCA Florida JFK Hospital, Atlantis, Florida
  - Nouvelle Clinical Research LLC, Cutler Bay, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward Health, Fort Lauderdale, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Baptist Health South Florida, Miami, Florida
  - NCA Research Institute - Florida, Naples, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Revival Clinical Research, Orlando, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Cleveland Clinic Foundation - Florida Weston Hospital, Weston, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - WellStar Health System, Inc, Marietta, Georgia
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Medical Group St. Vincent, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - MercyOne Iowa Heart, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kansas City Cardiac Arrhythmia Research LLC, Overland Park, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - University of Kentucky Research Foundation, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford St. John Hospital, Detroit, Michigan
  - Ascension Providence Hospital, Southfield, Michigan
  - Trinity health- Michigan Heart, Ypsilanti, Michigan
  - Minneapolis Heart Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota
  - North Mississippi Medical Center, Tupelo, Mississippi
  - St. Louis Heart and Vascular, Bridgeton, Missouri
  - St. Luke's Hospital, Chesterfield, Missouri
  - St. Lukes Hospital Kansas City (Mid America Heart Institute), Kansas City, Missouri
  - Bryan Heart, Lincoln, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Catholic Medical Center, Manchester, New Hampshire
  - Our Lady of Lourdes, Camden, New Jersey
  - Hackensack University Medical Center, Edison, New Jersey
  - Jersey Shore University Medical Center, Edison, New Jersey
  - Cooper Hospital- Cardiovascular Associates of Delaware Valley, Haddon Heights, New Jersey
  - Atlantic Health System- Morristown Medical Center, Morristown, New Jersey
  - Rutgers New Jersey Medical School, Piscataway, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Buffalo General, Buffalo, New York
  - Weill Cornell Medicine, New York, New York
  - Nuvance Health - Heart & Vascular Institute/Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - Nuvance Health - Vassar brothers Medical Center, Poughkeepsie, New York
  - Sanger Heart and Vascular, Charlotte, North Carolina
  - TriHealth Bethesda, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Mercy Health- St. Vincent Medical Center LLC, Toledo, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - St. Francis Hospital - Tulsa, Tulsa, Oklahoma
  - Providence Heart & Vascular, Portland, Oregon
  - Bryn Mawr Medical Specialists Association, Bryn Mawr, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - Penn State Hershey Medical City, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tower Health Reading Hospital, Reading, Pennsylvania
  - WellSpan Health, York, Pennsylvania
  - Prisma Health Upstate, Greenville, South Carolina
  - Bon Secours Upstate Cardiology, Greenville, South Carolina
  - North Central Heart, Sioux Falls, South Dakota
  - The Stern Cardiovascular Foundation, Germantown, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Ascension Seton, Austin, Texas
  - Austin Heart, Austin, Texas
  - Baylor Scott and White Research Institute, Dallas, Texas
  - HCA Medical City Dallas, Dallas, Texas
  - Baylor Scott White- All Saints- Fort Worth, Fort Worth, Texas
  - Medical City Fort Worth Hospital, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Heart Rhythm Specialists, McKinney, Texas
  - Baylor Scott and White- The Heart Hospital- Plano, Plano, Texas
  - Baylor Scott and White Research Institute - Round Rock, Round Rock, Texas
  - Methodist Hospital, San Antonio, Texas
  - Bon Secours St. Mary's, Richmond, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Peace Health, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abraham WT, Kuck KH, Goldsmith RL, Lindenfeld J, Reddy VY, Carson PE, Mann DL, Saville B, Parise H, Chan R, Wiegn P, Hastings JL, Kaplan AJ, Edelmann F, Luthje L, Kahwash R, Tomassoni GF, Gutterman DD, Stagg A, Burkhoff D, Hasenfuss G. A Randomized Controlled Trial to Evaluate the Safety and Efficacy of Cardiac Contractility Modulation. JACC Heart Fail. 2018 Oct;6(10):874-883. doi: 10.1016/j.jchf.2018.04.010. Epub 2018 May 10. PMID 29754812
- [Background] Wiegn P, Chan R, Jost C, Saville BR, Parise H, Prutchi D, Carson PE, Stagg A, Goldsmith RL, Burkhoff D. Safety, Performance, and Efficacy of Cardiac Contractility Modulation Delivered by the 2-Lead Optimizer Smart System: The FIX-HF-5C2 Study. Circ Heart Fail. 2020 Apr;13(4):e006512. doi: 10.1161/CIRCHEARTFAILURE.119.006512. Epub 2020 Apr 8. PMID 32264716
- [Background] Tschope C, Butler J, Farmakis D, Morley D, Rao I, Filippatos G. Clinical effects of cardiac contractility modulation in heart failure with mildly reduced systolic function. ESC Heart Fail. 2020 Dec;7(6):3531-3535. doi: 10.1002/ehf2.13126. Epub 2020 Dec 3. PMID 33274601
- [Background] Tschope C, Van Linthout S, Spillmann F, Klein O, Biewener S, Remppis A, Gutterman D, Linke WA, Pieske B, Hamdani N, Roser M. Cardiac contractility modulation signals improve exercise intolerance and maladaptive regulation of cardiac key proteins for systolic and diastolic function in HFpEF. Int J Cardiol. 2016 Jan 15;203:1061-6. doi: 10.1016/j.ijcard.2015.10.208. Epub 2015 Oct 27. No abstract available. PMID 26638055